CLINICAL TRIAL: NCT02295202
Title: Impact of Obstructive Sleep Apnea Treatment in Patients With Metabolic Syndrome: A Randomized Study
Brief Title: Impact of Obstructive Sleep Apnea Treatment in Patients With Metabolic Syndrome
Acronym: TREATOSA-MS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fleury (Unknown)
Responsible Party: Principal Investigator, Luciano F Drager, MD, PhD, Luciano F. Drager, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDC 4075/14/055
Record Dates: First submitted 2014-11-12; First posted 2014-11-20 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Sleep Apnea; Metabolic Syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes; Metabolic Syndrome | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Experimental): CPAP: Continuous Positive Airway Pressure - Device used for treating OSA during sleep.
  Interventions: Device: CPAP (REMstar System One Plus - Philips Medical Systems)
- Placebo (Placebo Comparator): Nasal Strips
  Interventions: Device: Nasal strips

INTERVENTIONS:
Device: CPAP (REMstar System One Plus - Philips Medical Systems) — Standard device for treating obstructive sleep apnea.
  Arms: CPAP
Device: Nasal strips
  Arms: Placebo

SUMMARY:
Obstructive Sleep Apnea (OSA) is a common condition that may induce hemodynamic and metabolic dysregulation. However, it is not clear if OSA is a mere epiphenomenon or contributes to increase the morbidity associated with metabolic syndrome. This study was designed to evaluate the impact of OSA treatment with CPAP in consecutive patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic Syndrome (ATP III)
* Moderate to severe OSA

Exclusion Criteria:

* Smokers
* Patients under chronic use of medications
* Neurological diseases
* Coronary artery disease
* Acute heart failure
* Chronic renal failure (GFR < 30 ml/min)
* Chronic obstructive pulmonary disease
* Mild OSA and patients with BMI over 40 kg/m2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03; Primary Completion 2019-04 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Reversibility of Metabolic Syndrome criteria | 6 months

SECONDARY OUTCOMES:
Abdominal fat | 6 months
  Abdominal CT
Hepatic steatosis | 6 months
  Abdominal CT
carotid intima-media thickness | 6 months
  Carotid ultrasound
endothelial function | 6 months
  Braquial artery ultrasound (flow mediated dilation, %)
coronary atherosclerosis | 6 months
  Coronary CT
Inflammatory markers | 6 months
  C-reactive protein
Metabolomics | 6 months
  Metabolomic analysis (intended to be a sub-study)
MicroRNAs | 6 months
  MicroRNAs analysis (intended to be a sub-study)
Epicardic fat | 6 months
  Epicardic fat quantification by CT (intended to be a sub-study)
Heart remodeling | 6 months
  Evaluated by Tranthoracic echocardiography (intended to be a sub-study)

CONTACTS AND LOCATIONS:
Overall Officials: Luciano F Drager, MD, PhD, Principal Investigator — Heart Institute (InCor), University of Sao Paulo Medical School
Locations (1):
- Luciano Drager, São Paulo, Brazil

REFERENCES:
- [Derived] Giampa SQC, Furlan SF, Freitas LS, Macedo TA, Lebkuchen A, Cardozo KHM, Carvalho VM, Martins FC, Azam IFB, Costa-Hong V, Lopes HF, Baptista ML, Rochitte CE, Bortolotto LA, Lorenzi-Filho G, Drager LF. Effects of CPAP on Metabolic Syndrome in Patients With OSA: A Randomized Trial. Chest. 2022 May;161(5):1370-1381. doi: 10.1016/j.chest.2021.12.669. Epub 2022 Jan 19. PMID 35063452